CLINICAL TRIAL: NCT00761332
Title: An Observational Study to Assess Back Pain in Patients With Severe Osteoporosis Treated With Teriparatide Versus Antiresorptives
Brief Title: Back Pain in Patients With Severe Osteoporosis
Status: Completed | Type: Observational
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Other Study IDs: 11837; B3D-CR-B013 (Other: Eli Lilly)
Record Dates: First submitted 2008-09-25; First posted 2008-09-29 (Estimated); Last update posted 2011-06-21 (Estimated); Status verified 2011-06

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Teriparatide; Raloxifene Hydrochloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Teriparatide: Patients treated with teriparatide
  Interventions: Drug: teriparatide
- Antiresorptive: Patients treated with antiresorptive therapy
  Interventions: Drug: antiresorptives

INTERVENTIONS:
Drug: teriparatide — treatment will be prescribed according to usual standard of care
  Other Names: Forteo; Forsteo; LY333334
  Groups: Teriparatide
Drug: antiresorptives — treatment will be prescribed according to usual standard of care
  Other Names: raloxifene, daily or weekly bisphosphonates
  Groups: Antiresorptive

SUMMARY:
The purpose of this study is to compare the effectiveness of teriparatide versus therapies that decrease bone loss to prevent new or worsening back pain in patients with osteoporosis seen in clinical practice.

DETAILED DESCRIPTION:
Study B3D-CR-B013 is a prospective observational study to compare changes in back pain among patients treated with teriparatide versus those treated with antiresorptives (raloxifene, daily or weekly bisphosphonates).

ELIGIBILITY:
Inclusion Criteria:

* Men and postmenopausal women who have a previous vertebral osteoporotic fracture that was sustained at least 6 weeks prior to joining the study.
* Patients who are free of severe or chronically disabling conditions other than osteoporosis.
* Patients who are not currently receiving and have not previously received teriparatide.
* Patients who agree to participate, return to follow-up visits, and who have signed informed consent to participate in the study.
* Patients, who in the opinion of the prescribing physician, are eligible to receive the intended treatment and comply with all the recommendations stated in the relevant product information.

Exclusion Criteria:

* Are investigator site personnel directly affiliated with the study and/or their immediate families. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
* Are Lilly employees (that is, employees, temporary contract workers, or designees responsible for conducting the study). Immediate family of Lilly employees may participate in Lilly-sponsored clinical trials, but are not permitted to participate at a Lilly facility.
* Patients who have any contraindications according to the relevant product information in the country in which they are being treated.
* Patients who are simultaneously participating in a different study that includes a treatment intervention and/or an investigational drug.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Routine clinical practice
Sampling Method: Non-Probability Sample
Enrollment: 650 (Actual)
Dates: Start 2008-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
New or worsening back pain as measured by a specific question in the Back Pain Questionnaire | 12 months

SECONDARY OUTCOMES:
Risk of developing moderate or severe back pain | 12 months
Changes in back pain severity using a Visual Analog Scale | 12 months
Treatment persistence, (days on therapy) | 12 months
Changes in health-related quality of life by completing the EuroQoL Scale (EQ-5D) | 12 months
Incidence of nontraumatic osteoporotic fractures | 12 months
Incidence of adverse events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (15):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pokfulam, Hong Kong
- India (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ahmedabad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gūrgaon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyderabaad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagpur
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Delhi
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., George Town, Malaysia
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara, Mexico
- Pakistan (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Islamabad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lahore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rawalpindi
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Singapore, Singapore
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Suwon, South Korea
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taichung, Taiwan
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bangkok, Thailand